CLINICAL TRIAL: NCT04638452
Title: Evaluation of Behavioural, Psychological and Physiological Responses in People With Autism Spectrum Disorder (ASD) During a Blood Test in Routine Care Practice
Brief Title: Evaluation of Behavioural Psycho & Physiological Responses in People With ASD During a Blood Test in Routine Care Practice
Acronym: AUTICOPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A00693-36
Record Dates: First submitted 2020-10-15; First posted 2020-11-20 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorders; behaviour; emotions; Physiological reactions; Psychological reactions
MeSH Terms: conditions — Autism Spectrum Disorder; Behavior | interventions — Videotape Recording; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Epidemiology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidemiology (Other): Video recording of face, body movements and physiological parameters (heart rate, conductance using a wireless watch) of the participants during the blood test Passing self and hetero questionnaires of temotion felt and perceived.
  Interventions: Behavioral: Video & movements recording; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Video & movements recording — Video recording of face, body movements and physiological parameters (heart rate, conductance using a wireless watch) of the participants during the blood test
Behavioral: Questionnaires — Passing self and hetero questionnaires of emotion felt and perceived.

SUMMARY:
The project is a prospective study designed to characterize behaviour and its psycho-physiological correlates of participants with ASD (children and adults) in comparison with subjects without ASD matched in age during blood test in common practice.

DETAILED DESCRIPTION:
The project is a prospective study designed to characterize behaviour and its psycho-physiological correlates of participants with ASD (children and adults) in comparison with subjects without ASD matched in age during blood test in common practice.

The aim is to analyse in an automated and standardised way video recording during a blood test performed as part of routine follow-up care for people presenting ASD (children and adults), qualitative data (type of emotion) and quantitative (intensity)

1. Emotional facial reactions
2. Behavioural reactions (video recording of participants' movements)
3. Physiological reactions (wireless smart watch worn on the wrist)
4. Psychological reactions (self and hetero questionaires) to characterize the signs of pain and anxiety associated with this situation)

ELIGIBILITY:
Inclusion Criteria:

All participants :

* Person over 6 years of age
* Person who consent to participate in the study
* Membership of the social security scheme
* Person who not received analgesic treatment that may interfere with pain perception
* Person with medical prescription for blood sample

Participants with ASD :

* Person with ASD diagnosis
* If applicable, legal authority consent to participate in the study

Exclusion Criteria:

All participants :

* Person with unstabilized drug therapy
* Person with acute or chronic pain
* Person with pathology or receiving a treatment which can have an impact in modification of the pain
* Person with oculomotor and/or neuro-motor disorders
* Pregnant or breastfeeding woman
* Person with deprivation of liberty
* Person who no consent to participate in the study or no consent to realised video recording

Participants without ASD :

* Protected adult
* Person with ASD diagnosis

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Facial expression during blood sample | through study completion, an average of 1 to 6 months
  Evaluation of facial expression during blood sample in people with ASD as compared to healthy people with Face reader, Noldus sofware.
Body movement during blood sample | through study completion, an average of 1 to 6 months
  Evaluation of body movement during blood sample in people with ASD as compared to healthy people with EMPATICA watch and Face, Legs, Activity, Cry, Consolabilty (FLACC) scale

SECONDARY OUTCOMES:
Evaluation of emotion felt by participants during blood sample | through study completion, an average of 1 to 6 months
  Evaluation of emotion felt by participants (anxiety, stress, pain, apprehension…) during blood sample with implified Scale for Assessing Pain in Dyscommunicatives People with Autism Spectrum Disorders (ESSDA) and Pain Assessment Grid - Intellectual Disability (GEDDI) scales

CONTACTS AND LOCATIONS:
Overall Officials: Anouck AMESTOY, MD, Study Director — Physician
Locations (1):
- Centre Hospitalier Charles PERRENS, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hilton CL, Harper JD, Kueker RH, Lang AR, Abbacchi AM, Todorov A, LaVesser PD. Sensory responsiveness as a predictor of social severity in children with high functioning autism spectrum disorders. J Autism Dev Disord. 2010 Aug;40(8):937-45. doi: 10.1007/s10803-010-0944-8. PMID 20108030
- [Result] Hirvikoski T, Mittendorfer-Rutz E, Boman M, Larsson H, Lichtenstein P, Bolte S. Premature mortality in autism spectrum disorder. Br J Psychiatry. 2016 Mar;208(3):232-8. doi: 10.1192/bjp.bp.114.160192. Epub 2015 Nov 5. PMID 26541693
- [Result] Breau LM, Camfield CS, McGrath PJ, Finley GA. The incidence of pain in children with severe cognitive impairments. Arch Pediatr Adolesc Med. 2003 Dec;157(12):1219-26. doi: 10.1001/archpedi.157.12.1219. PMID 14662579
- [Result] Breau LM, Camfield CS, McGrath PJ, Finley GA. Risk factors for pain in children with severe cognitive impairments. Dev Med Child Neurol. 2004 Jun;46(6):364-71. doi: 10.1017/s001216220400060x. PMID 15174527
- [Result] Dubois A, Rattaz C, Pry R, Baghdadli A. [Autism and pain - a literature review]. Pain Res Manag. 2010 Jul-Aug;15(4):245-53. doi: 10.1155/2010/749275. French. PMID 20808970
- [Result] Allely CS. Pain sensitivity and observer perception of pain in individuals with autistic spectrum disorder. ScientificWorldJournal. 2013 Jun 13;2013:916178. doi: 10.1155/2013/916178. Print 2013. PMID 23843740